CLINICAL TRIAL: NCT05555888
Title: A Prospective Phase II Trial of Immunotherapy Combined With Short-course Radiotherapy in Early Low Rectal Cancer
Brief Title: The Combination of Immunotherapy and Neoadjuvant Short-course Radiotherapy in Early Rectal Cancer
Acronym: TORCH-E
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2022-227-2945
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Early Low Rectal Cancer
MeSH Terms: interventions — spartalizumab; toripalimab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): A total of 34 patients will receive 5*5Gy short-course radiotherapy, followed by 4 cycles of CAPOX chemotherapy and PD-1 antibody, finally receive the TEM or TME surgery.
  Interventions: Drug: PD-1 antibody; Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Short-course radiotherapy

INTERVENTIONS:
Drug: PD-1 antibody — PD-1 antibody (Toripalimab): 240mg d1 q3w
  Other Names: Toripalimab
Drug: Capecitabine — Capecitabine: 1000mg/m2 d1-14 q3w
  Other Names: Xeloda
Drug: Oxaliplatin — Oxaliplatin: 130mg/m2 d1 q3w
Radiation: Short-course radiotherapy — Shor-course radiotherapy: 25Gy/5Fx

SUMMARY:
The study evaluates the combination of immunotherapy of PD-1 antibody and neoadjuvant short-course radiotherapy in early low rectal cancer. A total of 34 patients will receive 5*5Gy short-course radiotherapy, followed by 4 cycles of capecitabine plus oxaliplatin (CAPOX) chemotherapy and PD-1 antibody, finally receive the local excision(TEM) or total mesorectal excision (TME). The rate of complete response (cCR+pCR), Organ retention rate, long-term prognosis, and adverse effects will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-70 years old, female and male
2. pathological confirmed adenocarcinoma
3. clinical stage T1-3bN0, tumor maximum diameter less than 4cm
4. the distance from anal verge less than 5 cm
5. without distance metastases
6. KPS >=70
7. with good compliance
8. microsatellite repair status is MSS/pMMR
9. without previous anti-cancer therapy or immunotherapy
10. signed the inform consent

Exclusion Criteria:

1. pregnancy or breast-feeding women
2. pathological confirmed signet ring cell carcinoma
3. clinical stage T1N0 and can be resected locally
4. history of other malignancies within 5 years
5. serious medical illness, such as severe mental disorders, cardiac disease, uncontrolled infection, etc.
6. immunodeficiency disease or long-term using of immunosuppressive agents
7. baseline blood and biochemical indicators do not meet the following criteria: neutrophils≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L, ALT/AST ≤2.5 ULN, Cr≤ 1 ULN
8. DPD deficiency
9. allergic to any component of the therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) rate | The status of cCR will be evaluated after the completion of neoadjuvant therapy. The pCR rate will be evaluated after surgery. The cCR patients who adopted W&W strategy will be included into the CR rate caluculation.
  Rate of complete response (CR), including the rate of pathologic complete response (pCR) after surgery and the rate of cCR with W&W strategy.

SECONDARY OUTCOMES:
Organ preservation rate | from date of receiving neoadjuvant therapy, assessed up to 2 years
  Rate of patients who underwent organ preservation via WW or TEM after neoadjuvant therapy
Grade 3-4 adverse effects rate | From date of initiation of treatment until the date of death from any cause, assessed up to 5 years
  Rate of chemotherapy, radiotherapy and immunotherapy related adverse events
3 year disease free survival rate | From date of initiation of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  Rate of 3 year disease free survival
3 year local recurrence free survival rate | From date of initiation of treatment until the date of first documented pelvic failure, assessed up to 36 months.
  Rate of 3 year local recurrence free survival
3 year overall survival rate | From date of initiation of treatment until the date of death from any cause, assessed up to 36 months.
  Rate of 3 year overall survival
10 year Quality of Life | From date of initiation of treatment until the date of death from any cause, assessed up to 10 years
  Quality of life will be evaluated using EORTC QLQ-C30, EORTC QLQ-CR29, LARS score and Wexner score.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the related article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following related article publication.
Access Criteria: Proposals should be directed to xxx@yyy. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link will to be included).

REFERENCES:
- [Derived] Chen Y, Wang Y, Zhang H, Wan J, Shen L, Wang Y, Zhou M, Wu R, Yang W, Zhou S, Cai S, Li X, Zhang Z, Xia F. Short-course radiotherapy combined with chemotherapy and PD-1 inhibitor in low-lying early rectal cancer: study protocol for a single-arm, multicentre, prospective, phase II trial (TORCH-E). BMJ Open. 2023 Oct 6;13(10):e076048. doi: 10.1136/bmjopen-2023-076048. PMID 37802608